CLINICAL TRIAL: NCT04857450
Title: Anesthesia for Upper Endoscopy and Colonoscopy in Cardiac Patients With Acute Anemia: Pretreatment With Low-dose Ketamine Can Reduce the Dose of Etomidate. A Randomized Clinical Trial.
Brief Title: Anesthesia for Upper Endoscopy and Colonoscopy in Cardiac Patients With Acute Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mostafa Mohammed Elsaid Elhamamsy, Anesthesia Consultant, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E-20-4814
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Anemia; Cardiomyopathies; Pulmonary Hypertension
Keywords: Etomidate; Ketamine; Colonoscopy; Upper endoscopyPulmonary Hy
MeSH Terms: conditions — Anemia; Cardiomyopathies; Hypertension, Pulmonary | interventions — Etomidate; Ketamine

STUDY DESIGN:
Intervention Model Description: Sixty adult cardiac patients, older than 18 with ASA II or III physical status who underwent upper endoscopy together with colonoscopy for management of acute anemia in the cardiac intensive care units from November 2020 - October 2021. They were randomly divided into two groups. All patients received 0.05 mg/kg midazolam and 1µg/kg fentanyl slow IV as basal sedation and analgesia, then :
  Group (E): Received Etomidate 0.1 mg/kg IV over 20-30 seconds, followed by 0.05 mg/kg IV and repeated when needed, and Group (KE): Received Ketamine 0.5 mg/kg IV over 20-30 seconds followed by Etomidate 0.05 mg/kg IV over 20-30 seconds and repeated when needed.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants including care provider and outcome assessors will unaware of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Etomidate (Sham Comparator): Received Etomidate 0.2 mg/kg IV over 30 seconds, followed by 0.05 mg/kg IV and repeated when needed.
  Interventions: Drug: Etomidate
- Ketamine-Etomidate (Active Comparator): Received Ketamine 0.5 mg/kg IV over 30 seconds then Etomidate 0.1 mg/kg IV over 30 seconds, followed by 0.05 mg/kg IV and repeated when needed.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Etomidate — Received Etomidate 0.2 mg/kg IV over 30 seconds, followed by Etomidate 0.05 mg/kg IV and repeated when needed.
  Arms: Etomidate
Drug: Ketamine Hydrochloride — Received Ketamine 0.5 mg/kg IV over 30 seconds then Etomidate 0.1 mg/kg IV over 30 seconds, followed by 0.05 mg/kg IV and repeated when needed.
  Arms: Ketamine-Etomidate

SUMMARY:
The aim of this study was to try to reduce the required dose of etomidate used in anesthesia for upper endoscopy and colonoscopy in critically ill cardiac patients who complain of severe anemia in cardiac intensive care units by using a low dose of ketamine, which helps to reduce the side effects of etomidate, the most important of which is its suppressive effect on the adrenal gland and the secretion of cortisol in such critical cases, while maintaining hemodynamic stability, and the patient's satisfaction.

DETAILED DESCRIPTION:
This Prospective Randomized Clinical Trial will be done in the period from November 2020 - October 2021, after approval of our local ethical committee, and based upon written informed consent, included sixty cardiac patients, ASA physical statuses III or IV, admitted in CCU and SICU, and scheduled for upper endoscopy together with colonoscopy for diagnosis and management of acute anemia.

The study will be performed in the CCU or SICU with the presence of all emergency equipment's. The gastroenterologist who performed the colonoscopies will be blinded from the type of drugs used for sedation.

All patients will receive a colonic preparation protocol before the operation, and bowel cleansing will be performed, and all patients will be fasting 8 hours before the procedures.

Anesthesia management:

After establishment of IV access, standard monitoring will be performed (noninvasive blood pressure, ECG, SpO2, and BIS using (Masimo) monitor).

Nasal cannula for oxygen (6 l/min) will be connected to all patients, then midazolam 0.03mg/kg IV as a premedication, and fentanyl 1µg/kg IV will be injected to all patients.

By the means of sealed envelope technique, patients will be randomly divided into two groups:

Group (E): Received Etomidate 0.2 mg/kg IV over 30 seconds, followed by 0.05 mg/kg IV and repeated when needed.

Group (KE): Received Ketamine 0.5 mg/kg IV over 30 seconds then Etomidate 0.1 mg/kg IV over 30 seconds, followed by 0.05 mg/kg IV and repeated when needed.

The additional dose of etomidate will be determined by the anesthesiologist to achieve 4-5 sedation level of Ramsay Sedation Scale or BIS above 60.

Complications during procedure will be considered and defined as:

1. Hypotension: decrease of baseline systolic blood pressure (SBP) >30%, or decrease of baseline diastolic blood pressure (DBP) >30%, and this will be treated by phenylephrine 100-200 µg IV boluses.
2. Bradycardia: decrease of HR < 50/min, and this will be treated by atropine 0.5 mg IV boluses.
3. Apnea: spontaneous breathing > 30 sec, or SpO2 < 85%, and this will be treated by assisted manual ventilation using AMBU bag and face mask.

During the procedure the level of sedation will be assessed every five minutes after administration of anesthetic drugs using Ramsay Sedation Scale (RSS) [18]: (1 = Anxious or restless or both, 2 = Cooperative, 3 = Responding to commands, 4 = Brisk response to stimulus, 5 = Sluggish response to stimulus, 6 = No response to stimulus), in addition to BIS.

The use of standard monitoring will be continued until the patients were fully awake. At the end of the procedure, total etomidate dose, the duration of the procedure, and the recovery time of the patients were recorded.

After full recovery and when the patients are alert enough to express their attitude regarding the intra-procedural events, they will be asked to score their level of satisfaction during the procedure in terms of recalling any painful or other undesirable intra-procedural events.

Patient's satisfaction level willbe assessed with a Likert five-item scoring system [19]:

(1 = Not satisfied at all, 2 = slightly satisfied, 3 = somewhat satisfied, 4 = very satisfied, and 5 = extremely satisfied).

Serum cortisol before and 6 hours after the procedure will be estimated in this clinical trial to calculate the percentage of suppression in both groups.

Statistical Analysis:

Sample size was calculated using: Calculator.net Home / math / sample size calculator. Sample size of 30 cases in each group was calculated to have at least an 80% power to detect the expected differences between the two groups with respect to the primary goal.

Group comparison willbe performed between groups E and KE to analyze differences. Mean, standard deviation (SD), median, frequency, and percentage (%) will be used in the descriptive statistics of the quantitative and qualitative data. Mann-Whitney U test will be used in the analysis of quantitative independent data. Chi-square test will be used to analyze qualitative independent data, and Fischer's test will be used when chi-square test conditions were not met. For comparison of the sedation score data, hemodynamic parameters and SpO2 values, the repeated measurement analysis will be used. P value <0.05 will be considered statistically significant. SPSS v23.0 program will be used for all the analysis.

ELIGIBILITY:
Inclusion Criteria:

* - Age 18 - 65 years,
* ASA II-III
* Ejection fraction (EF) > 30%.

Exclusion Criteria:- Poor left ventricular function (ejection fraction < 30%).

* Recent myocardial infarction (last seven days),
* Patients with uncontrolled chronic disease (uncontrolled diabetes mellitus (DM) and hypertension),
* Known history of hypersensitivity to midazolam, fentanyl, etomidate, Or ketamine,
* Severe respiratory, hepatic or renal failure,
* History of neurological disorders or convulsions,
* In addition, any need for further anesthetic drug administration other than the study protocol was another exclusion criterion of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum cortisl level | From preoperative baseline to post operative after 6 hours
  Primary goal was to prove that if we combined etomidate with small dose of ketamine, the level of cortisol will be decreased to a lesser extent than in case we use etomidate alone. measurement will be done peoperative and 6 hours after the procedure

SECONDARY OUTCOMES:
Incidence of perioperative cardiopulmonary complications | From preoperative till postoperative 6 hours
  1. Hypotension: decrease of baseline systolic blood pressure (SBP) >30%, or decrease of baseline diastolic blood pressure (DBP) >30%, and this was treated by phenylephrine 100-200 µg IV boluses.
  2. Bradycardia: decrease of HR < 50/min, and this was treated by atropine 0.5 mg IV boluses.
  3. Apnea: spontaneous breathing > 30 sec, or SpO2 < 85%, and this was treated by assisted manual ventilation using AMBU bag and face mask.
Level of pateint satisfaction | From preoperative till full recovery after 6 hours
  After full recovery and when the patients were alert enough to express their attitude regarding the intra-procedural events, they will be asked to score their level of satisfaction during the procedure in terms of recalling any painful or other undesirable intra-procedural events.
  Patient's satisfaction level will be assessed with a Likert five-item scoring system :
  (1 = Not satisfied at all, 2 = slightly satisfied, 3 = somewhat satisfied, 4 = very satisfied, and 5 = extremely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Rubie M de Ocampo, Study Director — INSTITUTIONAL REVIEW BOARD King Saud University
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2022
Access Criteria: IPD data will be available on request through email.

REFERENCES:
- [Result] Corwin HL, Krantz SB. Anemia of the critically ill: "acute" anemia of chronic disease. Crit Care Med. 2000 Aug;28(8):3098-9. doi: 10.1097/00003246-200008000-00079. No abstract available. PMID 10966311
- [Result] van Leerdam ME, Vreeburg EM, Rauws EA, Geraedts AA, Tijssen JG, Reitsma JB, Tytgat GN. Acute upper GI bleeding: did anything change? Time trend analysis of incidence and outcome of acute upper GI bleeding between 1993/1994 and 2000. Am J Gastroenterol. 2003 Jul;98(7):1494-9. doi: 10.1111/j.1572-0241.2003.07517.x. PMID 12873568
- [Result] Colle I, Wilmer A, Le Moine O, Debruyne R, Delwaide J, Dhondt E, Macken E, Penaloza A, Piessevaux H, Stephenne X, Van Biervliet S, Laterre PF. Upper gastrointestinal tract bleeding management: Belgian guidelines for adults and children. Acta Gastroenterol Belg. 2011 Mar;74(1):45-66. PMID 21563653
- [Result] Regula J, Sokol-Kobielska E. Sedation in endoscopy: when and how. Best Pract Res Clin Gastroenterol. 2008;22(5):945-57. doi: 10.1016/j.bpg.2008.06.002. PMID 18790440
- [Result] Habibi MR, Baradari AG, Soleimani A, Emami Zeydi A, Nia HS, Habibi A, Onagh N. Hemodynamic responses to etomidate versus ketamine-thiopental sodium combination for anesthetic induction in coronary artery bypass graft surgery patients with low ejection fraction: a double-blind, randomized, clinical trial. J Clin Diagn Res. 2014 Oct;8(10):GC01-5. doi: 10.7860/JCDR/2014/10237.5006. Epub 2014 Oct 20. PMID 25478364
- [Result] Bovill JG. Intravenous anesthesia for the patient with left ventricular dysfunction. Semin Cardiothorac Vasc Anesth. 2006 Mar;10(1):43-8. doi: 10.1177/108925320601000108. PMID 16703233
- [Result] Forman SA. Clinical and molecular pharmacology of etomidate. Anesthesiology. 2011 Mar;114(3):695-707. doi: 10.1097/ALN.0b013e3181ff72b5. PMID 21263301
- [Result] Wanscher M, Tonnesen E, Huttel M, Larsen K. Etomidate infusion and adrenocortical function. A study in elective surgery. Acta Anaesthesiol Scand. 1985 Jul;29(5):483-5. doi: 10.1111/j.1399-6576.1985.tb02238.x. PMID 4036533
- [Result] Heidari SM, Loghmani P. Assessment of the effects of ketamine-fentanyl combination versus propofol-remifentanil combination for sedation during endoscopic retrograde cholangiopancreatography. J Res Med Sci. 2014 Sep;19(9):860-6. PMID 25535501
- [Result] Rai K, Hegde AM, Goel K. Sedation in uncooperative children undergoing dental procedures: a comparative evaluation of midazolam, propofol and ketamine. J Clin Pediatr Dent. 2007 Fall;32(1):1-4. doi: 10.17796/jcpd.32.1.v74872j8n74qu81k. PMID 18274461
- [Result] Zed PJ, Mabasa VH, Slavik RS, Abu-Laban RB. Etomidate for rapid sequence intubation in the emergency department: is adrenal suppression a concern? CJEM. 2006 Sep;8(5):347-50. doi: 10.1017/s1481803500014044. PMID 17338847
- [Result] Varga I, Racz K, Kiss R, Futo L, Toth M, Sergev O, Glaz E. Direct inhibitory effect of etomidate on corticosteroid secretion in human pathologic adrenocortical cells. Steroids. 1993 Feb;58(2):64-8. doi: 10.1016/0039-128x(93)90054-q. PMID 8387232
- [Result] Wu GN, Xu HJ, Liu FF, Wu X, Zhou H. Low-Dose Ketamine Pretreatment Reduces the Incidence and Severity of Myoclonus Induced by Etomidate: A Randomized, Double-Blinded, Controlled Clinical Trial. Medicine (Baltimore). 2016 Feb;95(6):e2701. doi: 10.1097/MD.0000000000002701. PMID 26871805
- [Derived] Elhamamsy MM, Aldemerdash AM, Zahran FB, Ezz GFM, AlSaud SA, Boules ML, Abdelhady MA, Hamed MA. Effects of adding low-dose ketamine to etomidate on serum cortisol levels in critically ill cardiac patients: a randomized clinical trial. BMC Anesthesiol. 2022 Apr 21;22(1):114. doi: 10.1186/s12871-022-01654-0. PMID 35448950